CLINICAL TRIAL: NCT05145231
Title: valıdıty and relıabılıty of the turkısh versıon of the functıonal mobılıty Scale ın ındıvıduals wıth Cerebral Palsy (Fms)
Brief Title: valıdıty and relıabılıty of the turkısh versıon of the functıonal mobılıty Scale ın ındıvıduals wıth Cerebral Palsy
Acronym: FMS
Status: Completed | Type: Observational
Sponsor: Nursena Güçlü (Other)
Collaborators: Kırıkkale University (Other)
Responsible Party: Sponsor-Investigator, Nursena Güçlü, physiotherapist, Kırıkkale University
Organization: Kırıkkale University (Other)
Other Study IDs: Kirikkaleüniversity3
Record Dates: First submitted 2021-10-01; First posted 2021-12-06 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy
Keywords: serebral palsi; GMFCS; Functional Mobility Scale; Abiloco-kids
MeSH Terms: conditions — Cerebral Palsy | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- grup 1: GMFCS PEDİ ABİLOCO-KİDS FMS
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — The scales will be filled by asking the family.

SUMMARY:
Cerebral palsy (CP) describes a group of persistent disorders in movement and postural development that cause activity limitation, attributed to non-progressive disturbances occurring in the developing fetal or infant brain.

Motor disorders of cerebral palsy are often accompanied by sensory, perception, cognition, communication and behavioral disorders due to epilepsy and secondary musculoskeletal problems.(Rosenbaum et al. 2007) Within the ICF, body functions are the physiological functions of body systems and anatomical parts of the body, such as body structures, organs, limbs, and components.

Disorders are problems that appear as a significant deviation or loss in body functions or structure. The primary injury in CP is a brain lesion resulting from an upper motor neuron lesion that is thought to have a number of positive and negative features. Positive traits include spasticity, hyperreflexia, and co-contraction, while negative traits include weakness, loss of selective motor control, and balance and coordination deficits.

The aim of the study is to examine the validity and reliability of the Turkish version of the Functional Mobility Scale (FMS) in individuals with cerebral palsy.

DETAILED DESCRIPTION:
GROSS MOTOR FUNCTİON CLASSİFİCATİON SYSTEM (GMFCS):

Level I: Walks without restrictions. Level II: Walks with restrictions. Level III: Walks using hand-held mobility devices. Level IV: Self-movement is limited. Can use a motorized mobility vehicle. Level V: Transported in a manual wheelchair. Differences Between Levels

Differences Between Levels I and II:

Compared to children/teens in Level I, children/teenagers in Level II have limitations in walking and balance. They may need hand-held mobility devices when they first learn to walk. They can use a wheeled mobility vehicle for long distance trips outside the home and in the community. They need the use of handrails when going up and down stairs. He does not have the ability to run and jump.

Differences Between Levels II and III:

Children and teenagers at Level II can walk without a hand-held mobility device after age 4 (although they prefer to use it occasionally). Children and youth in Level III use hand-held mobility devices to walk indoors and use wheeled mobility devices outside the home and in the community.

Differences Between Level III and IV:

Children and teenagers in Level III sit on their own or need very nervous external support to sit, are more independent in standing displacements, and walk with a hand-held mobility device. Children/teens at Level IV are functional seated (usually supported), but self-mobility is limited. Children and young people in Level IV are mostly transported in a manual wheelchair or use a motorized mobility vehicle.

Differences Between Levels IV and V:

Children and teenagers at Level V have severe limitations in bass and trunk control and need extensive technological and physical assistance. Self-mobility is gained only when the child/youth learns how to use a motorized wheelchair (2).

PEDİATRİC EVALUATİON OF DİSABİLİTY INVENTORY (PEDI):

Evaluates activities of daily living (self-care, mobility, social function) in children aged between 6 months and 7.5 years. PEDI is a comprehensive clinical assessment tool that assesses children's functional ability and performance. The first section, the Functional Skills Section, consists of 197 items and is a direct measurement of the child's functional abilities. In this section, the Self-Care subsection consists of 73 items, the Mobility subsection 59 and the Social Functions subsection 65 items. The child is given points as "0=cannot" and "1=can" for the items in this section. At the end of each subsection, the scores of that section are summed up and the functional skills (FB) total score is obtained by adding the scores of the subsections. The second and third sections evaluate the help and form of assistance from caregivers. It occurs in self-care, mobility, and social function items. Evaluation with the help of the caregiver is graded as independent, observation, minimum, moderate, maximum, complete. Adaptation evaluation is examined in 4 categories as no adaptation, adaptations for the child, rehabilitation tools and intensive adaptation. In this study, the mobility section will be used (3).

ABILOCO- KIDS:

It is a valid and reliable locomotion abilities scale defined on 10 items. ABILOCO-KIDS, which measures mobility, was translated into Turkish and applied. ABİLOCO-kids questionnaire consisting of ten questions was filled according to the information given by the parents. Questions are evaluated on a five-point scale. Impossible, difficult, easy, (unobserved activity). It can be applied to children aged 5 and over. (4)

FUNCTIONAL MOBILITY SCALE (FMS):

FMS classifies functional mobility in children with CP by grading the ability to walk at three specific distances, 5, 50, and 500 meters, according to the need for assistive devices. The scale includes various assistive devices such as wheelchairs, walkers, crutches and sticks, and also includes walking without the need for assistive devices. It uses a six-point ordinal scale (1-6) to rate the assistance needed at each distance reflecting distances from home, school, and community.

6 points, Independent on all surfaces. It does not use any walking aids or require the assistance of another person when walking on all surfaces, including uneven floors. (sidewalks etc. and in a crowded environment.)

5 points, Independent on flat surfaces. Does not use walking aids or need someone else's help. It needs handrails for stairs.

4 points, uses a cane (one or two). Walks without the help of another person.

3 points uses crutches without someone else's help.

2 points use walker without anyone else's help.

1 point, Uses a wheelchair. Can stop for transfers, take a few steps assisted by another person or using a walker.

C = Crawling: Child crawls (5m) to be able to move around the house.

N = not valid : For example, the child does not complete the distance ( 500 m ) .(1)

ELIGIBILITY:
Inclusion Criteria:

* 4 to 18 years of age
* Being diagnosed with cerebral palsy
* The GMFCS level was determined to be between I-IV.

Exclusion Criteria:

* The parent who will answer the form does not know Turkish.
* Performing orthopedic surgery and botulinum toxin injection in the previous six months.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 4-18 years diagnosed with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
functional mobility scale | 2 week
  6 points, Independent on all surfaces. It does not use any walking aids or require the assistance of another person when walking on all surfaces, including uneven floors. (sidewalks etc. and in a crowded environment.)
  5 points, Independent on flat surfaces. Does not use walking aids or need someone else's help. It needs handrails for stairs.
  4 points, uses a cane (one or two). Walks without the help of another person.
  3 points uses crutches without someone else's help.
  2 points use walker without anyone else's help.
  1 point, Uses a wheelchair. Can stop for transfers, take a few steps assisted by another person or using a walker.
  C = Crawling: Child crawls (5m) to be able to move around the house.
  N = not valid : For example the child does not complete the distance ( 500 m ) .

CONTACTS AND LOCATIONS:
Overall Officials: saniye arslan, Study Director — kırıkkale üniversitesi
Locations (1):
- Yeni Kurtuluş Özel Eğitim Ve Rehabilitasyon Merkezi, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No